CLINICAL TRIAL: NCT04100746
Title: Treatment of Post Traumatic Asymmetrical Ankle Arthritis Using Low Tibial Osteotomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed sayed kamel, Resident in assiut university, Assiut University
Other Study IDs: ankle osteoarthritis
Record Dates: First submitted 2019-09-21; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Ankle Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: supramalleolar osteotomy — surgical intervention by using low tibial osteotomy
  Other Names: fibular osteotomy

SUMMARY:
Evaluation of joint preserving procedure for asymmetrical ankle arthritis regarding the improvement of alignment and its effect on symptoms

DETAILED DESCRIPTION:
The most common cause of end-stage ankle arthritis is trauma. Post traumatic ankle arthritis is accepted as the most common cause of ankle arthritis,with reports ranging from 70% to 80% of all ankle arthritis. Factors contributing to the development of posttraumatic ankle arthritis are the initial cartilage damage, malreduction ,nonunion, infections, and instability. In a retrospective study,found that 55% of patients with posttraumatic ankle arthritis presented with a varus malalignment, whereas 8% had valgus malalignment 1. Nonoperative treatments, including orthotics, wedges, shoe modifications,anti-inflammatory medications, and activity modification,are usually not successful. Although the gold standard treatment for ankle arthrosis remains ankle arthrodesis, the significant loss of motion in the ankle is limiting and may lead to the development of arthritis in adjacent joints in the hind foot and forefoot . Total ankle replacements (TAR) used only in older, low-demand patients with neutral alignment and intact stabilizing ligaments. Ankle arthroscopy is indicated in acute, recurring-acute, and chronic ankle pain to detect the possible presence of anterior ankle impingement (bony or soft tissue), syndesmotic injury, osteochondral defects and loose bodies . Supramalleolar osteotomy have been used for varus and valgus as well as sagittal and rotational deformities .Fibular osteotomy, Calcaneal slide osteotomy and osteotomies of the medial arch can be also used as joint preserving procedure. Our study is designed for evaluation of the effect of joint preserving procedures in young patient with asymmetrical ankle arthritis.

ELIGIBILITY:
Inclusion Criteria:

* 1-Age 18-60 years. 2-Symptomatic ankle osteoarthritis varus or valgus ankle deformity on X-ray with asymmetrical ankle arthritis.

  3-Patient had failure of conservative treatment. 4-Patient with clinical symptoms,such as pain with walking and limitation of daily and recreational activities.

Exclusion Criteria:

* 1- End-stage arthritis 2- Severe hindfoot instability that cannot be stabilized 3- Severe vascular or neurologic deficiency in the affected extremity 4 - Neuropathic disorders (eg, Charcot foot). 5- Diabetes,chronic liver disease,renal failure 6- Smoking, and rheumatic disease. 7- Condition altered bone quality (due to medication, large cysts,osteoporosis and osteopenia )

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patient with post traumatic ankle arthritis.Age 18-60 years.Symptomatic ankle OA with varus or valgus ankle deformity on X-ray with asymmetrical ankle arthritis.-Patient with clinical symptoms,such as pain with walking and limitation of daily and recreational activities.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
AOFAS score | one year
  Score measures of pain ,alignment,

SECONDARY OUTCOMES:
UNION Rate | 6 month
  union rate of supramalleolar osteotomy

CONTACTS AND LOCATIONS:
Overall Officials: fasil fahmy adam, prof, Principal Investigator — assiut university orthopedic and traumatology department

REFERENCES:
- [Background] Martin RL, Stewart GW, Conti SF. Posttraumatic ankle arthritis: an update on conservative and surgical management. J Orthop Sports Phys Ther. 2007 May;37(5):253-9. doi: 10.2519/jospt.2007.2404. PMID 17549954